CLINICAL TRIAL: NCT01184976
Title: Phase I, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity in Healthy Adult Males of a DNA Plasmid Vaccine for HS Avian Influenza (VGX-3400) Administered by Intramuscular (IM) Injection Followed by Electroporation (EP)
Brief Title: Study Of VGX-3400, H5N1 Avian Flu Virus Plasmid DNA With Electroporation Device In Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLU-001
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: H5N1; Avian Influenza; DNA Vaccine; Electroporation; Intramuscular (IM) Injection
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.6mg DNA/dose (Experimental): Subjects will receive a 2 dose series of VGX-3400 containing 0.6mg DNA/dose administered via IM injection + electroporation at Day 0 and Month 1
  Interventions: Biological: VGX-3400
- 2mg DNA/dose (Experimental): Subjects will receive a 2 dose series of VGX-3400 containing 2mg DNA/dose administered via IM injection + electroporation at Day 0 and Month 1
  Interventions: Biological: VGX-3400
- 6mg DNA/dose (Experimental): Subjects will receive a 2 dose series of VGX-3400 containing 6mg DNA/dose administered via IM injection + electroporation at Day 0 and Month 1
  Interventions: Biological: VGX-3400

INTERVENTIONS:
Biological: VGX-3400 — Plasmid DNA delivered via IM injection with electroporation

SUMMARY:
Research Hypothesis: VGX-3400 (DNA plasmids encoding the hemagglutinin (HA), neuraminidase (NA), and M2e-NP antigen of the H5N1 avian influenza virus) administered to healthy adult males by IM injection followed by EP will be generally well tolerated and immunogenic.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines. If required by local law, candidates must also authorize the release and use of protected health information (PHI)
* Male subjects 20-39 years of age
* Healthy subjects as judged by the Investigator based on medical history, physical examination, and normal results for an ECG, CBC, serum chemistries, CPK and urinalysis done up to 30 days prior to enrollment and administration of study drug
* Current nonsmoker
* Body mass index (BMI) ≤30 kg/m2
* Able and willing to comply with all study procedures.

Exclusion Criteria:

* Positive serological test for HIV virus, hepatitis C virus or hepatitis B virus surface antigen (HBsAg);
* Any concurrent condition requiring the continued use of systemic or topical steroids (excluding inhaled and eye drop-containing corticosteroids); or the use of immunosuppressive or immune modifying agents within 3 months prior to Day 0 other than corticosteroids; or systemic or topical corticosteroids which must be discontinued > 4 weeks prior to Day 0
* Administration of any blood product within 3 months of enrollment
* Prior receipt of an H5N1 influenza vaccine at any time
* Administration of any non-study vaccine in the 6 weeks prior to study enrollment
* Subject is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent;
* Metal implants at the site of injection, however, metal implants elsewhere are permitted and do not represent an exclusion criterion;
* Active substance abuse or use of drugs such as heroin, cocaine or other drugs of addiction or daily use of alcohol greater than 100 ml of whiskey or other liquor, greater than 300 ml of wine, or greater than 360 ml of beer daily during the study period or in the week prior to starting the study;
* Subjects whose deltoid or quadriceps is not available;
* Subjects receiving anti-viral drugs & with primary thrombocytopenia;
* Serious Adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain (Not excluded: a participant who had a non-anaphylactic adverse reaction to pertussis vaccine as a child);
* Autoimmune disease, including Guillain-Barré syndrome;
* Clinically significant medical condition, physical exam findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response;
  * A process that would require medication that affects the immune response;
  * Any contraindication to repeated injections or blood draws;
  * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period;
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or;
  * Any condition specifically listed among the exclusion criteria.
* Subjects with known prior illness or who is at risk for H5N1 Influenza A virus infection, i.e. exposure in the two weeks prior to study Day 0 to a person with known H5N1 Influenza virus infection or travel in the 2 weeks prior to Day 0 or during the course of the study to a region with known current cases of H5N1 Influenza virus infection;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
* Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Day 0 through Month 4
  Frequency, severity of local and systemic reactogenicity signs and symptoms, adverse events and serious adverse events

SECONDARY OUTCOMES:
Humoral and cellular Immune Responses | Day 0 through Month 4
  Values of antibody and cell-mediated immune responses to HA, NA and M2e-NP proteins

CONTACTS AND LOCATIONS:
Overall Officials: Minja Kim, Principal Investigator — Korea Univ. MC; Minsoo Park, Principal Investigator — Severance Hospital
Locations (2):
- South Korea (2):
  - Yonsei University Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul